CLINICAL TRIAL: NCT02754193
Title: Effects of Induced Moderate HYPOthermia on Mortality in Cardiogenic Shock Patients Rescued by Veno-arterial ExtraCorporeal Membrane Oxygenation (ECMO)
Acronym: HYPO-ECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A00377-44
Record Dates: First submitted 2016-04-12; First posted 2016-04-28 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-03

CONDITIONS: Cardiogenic Shock
Keywords: Venous-Arterial ExtraCorporeal Membrane Oxygenation
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate hypothermia (Experimental): Moderate hypothermia :Patients with cardiogenic shock treated with arteriovenous ECMO to a strategy of moderate hypothermia during 24 hours (Temperature at 33°C≤ T°C ≤34°C) associated with usual care
  Interventions: Other: moderate hypothermia
- Normothermia (No Intervention): Normothermia: Patients with cardiogenic shock treated with arteriovenous ECMO to a strategy of normothermia (36°C≤ T°C ≤37°C) associated with usual care

INTERVENTIONS:
Other: moderate hypothermia — moderate hypothermia will be induced using the heat controller of the VA-ECMO circuit. Temperature will be maintained between 33°C≤ T°C ≤34°C during 24 hours ± 1h followed by a progressive reheating (0.2±0.1°C/h) to reach 37 °C. Temperature at 37°C ± 0.3°C will be maintained during 48 hours ± 4h after having reached 37 °C.
  Arms: Moderate hypothermia

SUMMARY:
A multicenter, prospective, controlled, randomized (moderate hypothermia 33°C≤ T°C ≤34°C) during 24 hours ± 1h versus normothermia (36°C≤ T°C ≤37°C), comparative open trial will be conducted on two parallel groups of patients with cardiogenic shock treated with VA-ECMO.

The HYPO-ECMO trial will test the hypothesis that moderate hypothermia (temperature between 33°C≤ T°C ≤34°C) associated with VA-ECMO support results in a reduction in 30-day mortality in comparison with the normothermia group (36°C≤ T°C ≤37°C).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Intubated patients with cardiogenic shock treated with VA-ECMO
* Patient affiliated to social security plan

Exclusion Criteria:

* VA-ECMO after cardiac surgery for heart transplantation or lung transplantation or left or biventricular assist device implantation
* VA-ECMO for acute poisoning with cardio-toxic drugs
* Pregnancy
* Uncontrolled bleeding (bleeding despite medical intervention (surgery or drugs))
* Implantation of VA ECMO under cardiac massage with a duration of cardiac massage >45minutes
* Out of hospital refractory cardiac arrest
* Cerebral deficit with fixed dilated pupils
* Participation in another interventional research involving therapeutic modifications
* Patient moribund on the day of randomization
* Irreversible neurological pathology
* Minor patients
* Patients under tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
All-cause Mortality | Day 30
  The study objective is to determine whether early moderate hypothermia (33°C≤ T°C ≤34°C) is superior to normothermia (37°C ± 0.3°C) in patients with cardiogenic shock treated with VA-ECMO with respect to 30-day mortality

SECONDARY OUTCOMES:
All-cause mortality | Hour 48, Day 7, Day 60, day 180
  Evaluation of the impact of moderate hypothermia on mortality during hospitalization and up to 180 days
Venous Arterial ECMO duration | up to 180 days (from date of randomization until ECMO weaning)
  Evaluation of the impact of moderate hypothermia on VA-ECMO weaning time
Death | day 30, Day 60, Day 180
  Evaluation of the impact of moderate hypothermia on adverse cardiovascular events. Composite endpoint of death, cardiac transplant, escalation to Left Ventricular Assist Device, stroke (cf secondary outcome n° 4, 5;6;7)
cardiac transplant | day 30, Day 60, Day 180
  Evaluation of the impact of moderate hypothermia on adverse cardiovascular events. Composite endpoint of death, cardiac transplant, escalation to Left Ventricular Assist Device, stroke (cf secondary outcome n° 4, 5;6;7)
escalation to Left Ventricular Assist Device | day 30, Day 60, Day180
  Evaluation of the impact of moderate hypothermia on adverse cardiovascular events. Composite endpoint of death, cardiac transplant, escalation to Left Ventricular Assist Device, stroke (cf secondary outcome n° 4, 5;6;7)
Stroke | Day 30, Day 60, Day 180
  Evaluation of the impact of moderate hypothermia on adverse cardiovascular events. Composite endpoint of death, cardiac transplant, escalation to Left Ventricular Assist Device, stroke (cf secondary outcome n° 4, 5;6;7)
Cumulated amount of administered fluids | up to 180 days (from date of randomization until ECMO weaning)
  Evaluation of the impact of moderate hypothermia on necessity of fluid
Cumulated amount of vasopressors use | up to 180 days (from date of randomization until ECMO weaning)
  Evaluation of the impact of moderate hypothermia on necessity of vasopressor (norepinephrine, epinephrine)
Lactate | up to 180 days (from date of randomization until ECMO weaning)
  Evaluation of the impact of moderate hypothermia on lactate clearance
SOFA score | from baseline until Day 30
  Evaluation of the impact of moderate hypothermia on duration of organ failure
Mechanical ventilation | baseline, day 30, day 60 and day 180
  Evaluation of the impact of moderate hypothermia on mechanical ventilation support use
Renal replacement therapy | from baseline until day 30, day 60, day 180
  Evaluation of the impact of moderate hypothermia on renal replacement therapy use
Intensive care unit stay | Day 30; Day 60; Day 180
  Evaluation of the impact of moderate hypothermia on duration of ICU stay
hospitalization stay | Day 30; Day 60; Day 180
  Evaluation of the impact of moderate hypothermia on duration of total hospitalization
bleeding complications | Hour 48, Day 7
  Evaluation of the impact of moderate hypothermia on the risk of bleeding under ECMO
packed red blood cells transfused | Hour 48, Day 7
  Evaluation of the impact of moderate hypothermia on the risk of bleeding under ECMO
Infection | Hour 48, Day 7, Day 30, Day 60, day 180
  Evaluation of the impact of moderate hypothermia on risk of sepsis (pulmonary, blood, venous lines, cannulaes)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LEVY, Pr, Principal Investigator — CHRU Nancy; Alain COMBES, Pr, Study Chair — APHP-Pitié Salpêtrière; Fabrice VANHUYSE, Dr, Study Chair — CHRU Nancy; Nicolas GIRERD, Pr, Study Chair — CHRU Nancy; Patrick ROSSIGNOL, Pr, Study Chair — CHRU Nancy
Locations (20):
- France (20):
  - CHU Amiens - Picardie -Site sud, Amiens
  - CH Annecy Centre Hospitalier, Annecy
  - CHU Besançon Hôpital Jean Minjoz, Besançon
  - CHU Bordeaux - Groupe Hospitalier SaintAndré, Bordeaux
  - CHU Clermont-Ferrand -Hopital G. Montpied, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHU Lyon - Hôpital Louis Pradel, Lyon
  - APHM-Hôpital, de la Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes/ Hôpital Nord Laennec, Nantes
  - APHP- Hôpital Bichat, Paris
  - APHP- la Pitié Sapêtrière, Paris
  - Aphp-Hegp, Paris
  - APHP-Pitié, Paris
  - CHU Rennes Hôpital Pontchaillou, Rennes
  - Chu Rouen, Rouen
  - CHRU Strasbourg, Strasbourg
  - CHU Strasbourg/ NHC, Strasbourg
  - CHU Toulouse Hôpital - Pierre Paul Riquet, Toulouse
  - CHRU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baudry G, Girerd N, Duarte K, Monzo L, Delmas C, Van Spall HGC, Kimmoun A, Levy B. Sex-Related Prognosis of VA-ECMO-Treated Cardiogenic Shock: A Post Hoc Analysis of the HYPO-ECMO Trial. Circ Heart Fail. 2025 Aug;18(8):e012702. doi: 10.1161/CIRCHEARTFAILURE.124.012702. Epub 2025 May 20. PMID 40390595
- [Derived] Baudry G, Levy B, Duarte K, Monzo L, Combes A, Kimmoun A, Girerd N. Prognosis of refractory cardiogenic shock in de-novo versus acute-on-chronic heart failure: Insights from the HYPO-ECMO trial. J Crit Care. 2025 Jun;87:155043. doi: 10.1016/j.jcrc.2025.155043. Epub 2025 Feb 28. PMID 40023081
- [Derived] Levy B, Girerd N, Baudry G, Duarte K, Cuau S, Bakker J, Kimmoun A; HYPO-ECMO trial group and the International ECMO Network (ECMONet). Serial daily lactate levels association with 30-day outcome in cardiogenic shock patients treated with VA-ECMO: a post-hoc analysis of the HYPO-ECMO study. Ann Intensive Care. 2024 Mar 27;14(1):43. doi: 10.1186/s13613-024-01266-6. PMID 38536534
- [Derived] Levy B, Girerd N, Amour J, Besnier E, Nesseler N, Helms J, Delmas C, Sonneville R, Guidon C, Rozec B, David H, Bougon D, Chaouch O, Walid O, Herve D, Belin N, Gaide-Chevronnay L, Rossignol P, Kimmoun A, Duarte K, Slutsky AS, Brodie D, Fellahi JL, Ouattara A, Combes A; HYPO-ECMO Trial Group and the International ECMO Network (ECMONet). Effect of Moderate Hypothermia vs Normothermia on 30-Day Mortality in Patients With Cardiogenic Shock Receiving Venoarterial Extracorporeal Membrane Oxygenation: A Randomized Clinical Trial. JAMA. 2022 Feb 1;327(5):442-453. doi: 10.1001/jama.2021.24776. PMID 35103766
- [Derived] Jacquot A, Lepage X, Merckle L, Girerd N, Levy B. Protocol for a multicentre randomised controlled trial evaluating the effects of moderate hypothermia versus normothermia on mortality in patients with refractory cardiogenic shock rescued by venoarterial extracorporeal membrane oxygenation (VA-ECMO) (HYPO-ECMO study). BMJ Open. 2019 Oct 14;9(10):e031697. doi: 10.1136/bmjopen-2019-031697. PMID 31615800
- See also: Statistical analysis plan — https://cic-p-nancy.fr/wp-content/uploads/2021/01/HYPO-ECMO-SAP-2021.pdf